CLINICAL TRIAL: NCT02784366
Title: GI Complications in Cancer Immunotherapy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Michael Dougan, Attending physician, Massachusetts General Hospital
Other Study IDs: 15302
Record Dates: First submitted 2016-05-06; First posted 2016-05-27 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Malignant Melanoma
Keywords: Cancer immunotherapy; Ipilimumab
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool samples will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cancer immunotherapy patients - no GI side effect: Cancer immunotherapy patients who do not develop GI side effects.
- Cancer immunotherapy patients - develop GI side effects: Cancer immunotherapy patients who develop GI side effects

SUMMARY:
The purpose of this study is to establish a prospective observational cohort of cancer immunotherapy patients with GI side effects in order to identify biomarkers that predict GI complications due to treatment.

DETAILED DESCRIPTION:
Primary objective

* To create a data and bio-specimen repository to enhance both safety and efficacy of immunotherapy

Secondary objective

* Identify biomarkers that may predict GI toxicity in cancer patients undergoing immunotherapy
* Define the clinical course of intestinal inflammation and identify genetic factors of therapeutic response to GI medications
* Analyze genotype-phenotype correlations in GI side effects in patients undergoing cancer immunotherapy

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cancer
* Currently undergoing or have undergone immunotherapy

Exclusion Criteria:

* History of a total colectomy
* History of inflammatory bowel disease (either ulcerative colitis or Crohn's disease)
* History of colitis on chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of cancer who have undergone or will be undergoing immunotherapy will be eligible for recruitment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
GI disease activity | 12 weeks
  To evaluate GI disease activity associated with cancer immunotherapy through a series of standardized questionnaires that measure severity of GI symptoms.
Biospecimen collection | 12 weeks
  To collect stool, blood, and colon biopsies and have the ability to identify predictive biomarkers in patients that develop colitis as a result of cancer immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dougan, MD, PhD, Principal Investigator — Massachusetts General Hospital; Ryan J Sullivan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes